CLINICAL TRIAL: NCT02667093
Title: Bone Marrow and Peripheral Blood (PB) Samples From Patients With Leukemia and PB From Their BM Donors (BMD) to Identify Leukemia-Specific Antigens (LSA) and Graft Versus Host Disease Antigens (GVHDA) for Use in Cellular Immunotherapy
Brief Title: Samples From Leukemia Patients and Their Donors to Identify Specific Antigens
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: PersImmune, Inc (Industry)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Other Study IDs: Persimmune Sample Collection
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Leukemia; Acute Myeloid Leukemia; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples will be shipped to Persimmune for processing and storage with results shared with Dr. Ball and his lab at UCSD.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this project is to develop a process to identify highly personalized antigens that are uniquely expressed by the patient's own leukemia cells that can be used for cellular immune therapy.

DETAILED DESCRIPTION:
It is well known that tumor cells and leukemia cells express different surface structures (called antigens) that can serve as targets for cancer cell destruction by the immune system. Effective immune therapies are characterized by high specificity and low toxicity. One of the major obstacles impeding the use of these therapies as standard of care is the identification of good target antigens. In acute myeloid leukemia (AML) there is major patient to patient variation in leukemia antigens, so there is no universal AML cell target. Rather, each patient has a unique array of potential cell targets. Thanks to the rapid progress of new DNA/RNA sequencing technologies, the identification of these unique, patient-specific leukemia cell antigen-targets is now possible.

The purpose of this project is to develop a process to identify highly personalized antigens that are uniquely expressed by the patient's own leukemia cells that can be used for cellular immune therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML with plan to receive a bone marrow transplant

Exclusion Criteria:

* NA

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with leukemia and their potential bone marrow donors.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Genomics of patients with leukemia and their HLA matched bone marrow transplant donors. | 5 years
  To sequence the exome and transcriptome obtained from leukemia cells and the exome from their lymphocytes, and the lymphocytes from their HLA matched marrow transplant donors.

SECONDARY OUTCOMES:
Identification of patients' leukemia cell mutations and polymorphisms that are different from their HLA matched bone marrow transplant donors | 5 years
  To select leukemia specific mutations (aka, variants), ie those that are different from both the patient's non-leukemic cells and their HLA matched marrow transplant donor's immune cells by comparing Leukemia cell, Patient normal cell, and Donor exome sequences.
Immunogenic mutant neoantigen peptide selection | 5 years
  To select peptides that represent the sequences obtained from Aim 2, according to their ability to bind to the identical patient/donor T cell major histocompatibility receptors.
Peptide immunogenicity confirmation and donor T cell stimulation | 5 years
  To test the peptides from Aim 3 for their in vitro immunogenicity for T lymphocytes obtained from the donor.
Data analysis and interpretation | 5 years
  To create and analyze a database summarizing the data obtained from Aims 1-4 for the purpose of IND submission and clinical trial design.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Ball, MD, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - University of California San Diego, La Jolla, California
  - Northside Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Montagna D, Maccario R, Locatelli F, Rosti V, Yang Y, Farness P, Moretta A, Comoli P, Montini E, Vitiello A. Ex vivo priming for long-term maintenance of antileukemia human cytotoxic T cells suggests a general procedure for adoptive immunotherapy. Blood. 2001 Dec 1;98(12):3359-66. doi: 10.1182/blood.v98.12.3359. PMID 11719375
- [Background] Kreiter S, Castle JC, Tureci O, Sahin U. Targeting the tumor mutanome for personalized vaccination therapy. Oncoimmunology. 2012 Aug 1;1(5):768-769. doi: 10.4161/onci.19727. PMID 22934277
- [Background] Klebanoff CA, Gattinoni L, Restifo NP. Sorting through subsets: which T-cell populations mediate highly effective adoptive immunotherapy? J Immunother. 2012 Nov-Dec;35(9):651-60. doi: 10.1097/CJI.0b013e31827806e6. PMID 23090074
- [Background] Brenner MK. Will T-cell therapy for cancer ever be a standard of care? Cancer Gene Ther. 2012 Dec;19(12):818-21. doi: 10.1038/cgt.2012.74. Epub 2012 Oct 12. PMID 23059871